CLINICAL TRIAL: NCT06482073
Title: Molecular Analysis of Suspected or High-Risk Lung Cancer to Drive Individualized Care (Interception for Suspected Lung Cancer)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-000609; NCI-2024-04855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000609 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Lung Carcinoma; Metastatic Malignant Neoplasm in the Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients receive genomic counseling and genomic testing education, undergo blood or saliva collection, provide previously collected tissue sample and have medical records reviewed on study. Patients and healthcare providers receive results of any genetic variants found on testing.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the effectiveness of robotic biopsies in providing information about hereditary or cancer specific genetic variants that may have a role in diagnosis of cancer and to develop genetic results and medical record databank for future studies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assessing whether the percentage of samples adequate for WES (Whole Exome Sequencing)/WT (Wild-Type) sequencing is at least 80%.

II. Development of a data bank of WES/WT and germline sequencing data for future analyses.

OUTLINE: This is an observational study.

Patients receive genomic counseling and genomic testing education, undergo blood or saliva collection, provide previously collected tissue sample and have medical records reviewed on study. Patients and healthcare providers receive results of any genetic variants found on testing.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 18 years and older
* Subject is scheduled/was scheduled for a bronchoscopy as part of standard of care
* Subject with a moderate to high risk of lung cancer based on clinical demographic and radiologic information or with suspected metastatic disease
* Ability to provide blood or saliva sample
* Ability to provide archived tissue
* Subject is able to understand and adhere to study requirements and able to provide informed consent

Exclusion Criteria:

* Individuals who have situations that would limit compliance with the study requirements
* Institutionalized (i.e. federal medical prison)
* Pregnant
* Prior germline genetic testing with a 40+ multi-gene panel within the last 1 year of enrollment
* Prior somatic tissue (250+ gene) testing within the prior 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a bronchoscopy recruited through Mayo Clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Percent of samples adequate for sequencing | Up to 2 years
  Assessed based on the number of tissue samples determined to be adequate for WES (Whole Exome Sequencing)/WT (wild-type) sequencing.

SECONDARY OUTCOMES:
Data bank of genomic data | Up to 2 years
  A data bank of genomic data will be developed for future analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Janani S. Reisenauer, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials